CLINICAL TRIAL: NCT06819254
Title: Pilot Study of Fisetin to Improve Fatigue Among Older Adult Cancer Survivors
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: The Ambrose Monell Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB00125637
Record Dates: First submitted 2025-01-27; First posted 2025-02-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Fatigue
Keywords: cancer survivor; supplement; Fisetin
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: 1:1 randomization, cross-over design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fisetin - Placebo (Experimental): Two-week regimen of Fisetin supplement followed by two-week regimen of placebo.
  Interventions: Drug: Fisetin followed by Placebo
- Placebo - Fisetin (Experimental): Two-week regimen of placebo followed by two-week regimen of Fisetin supplement.
  Interventions: Drug: Placebo followed by Fisetin

INTERVENTIONS:
Drug: Fisetin followed by Placebo — Fisetin 20 mg/kg per dose twice daily on two consecutive days for two consecutive weeks. Participants will return on day 14 for a blood draw followed by a 14-day wash-out. At the 4-week visit participants will receive a cross-over placebo-controlled dosing regimen to be taken twice daily on two consecutive days for two consecutive weeks.
  Arms: Fisetin - Placebo
Drug: Placebo followed by Fisetin — Placebo twice daily on two consecutive days for two consecutive weeks. Participants will return on day 14 for a blood draw followed by a 14-day wash-out. At the 4-week visit participants will receive a cross-over Fisetin 20 mg/kg per dose twice daily on two consecutive days for two consecutive weeks.
  Arms: Placebo - Fisetin

SUMMARY:
The purpose of this study is to find out if taking a Fisetin supplement can decrease fatigue among older cancer survivors.

DETAILED DESCRIPTION:
Prospective double-blind placebo controlled, 14-day cross-over trial of patients aged 65 and over with a history of cancer with self-reported fatigue. Participants will be randomized and provided with Fisetin pills or placebo to take twice daily on two consecutive days for two consecutive weeks. Participants will return on day 14 for a blood draw followed by a 14 day wash-out. At the four-week visit participants will receive a cross-over placebo-controlled dosing regimen over two weeks. Follow-up phone calls for safety assessment and adherence review will occur at weeks 1 and 5. Follow-up assessments will be completed at 2, 4 and 6 weeks, and a post-treatment phone call assessment completed at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported history of cancer diagnosed > 12 months prior to enrollment excluding non-melanoma skin cancer with no evidence of disease at enrollment.
* Eligible solid tumor cancer types include Stage 1-3 breast, lung, head and neck, colorectal, anal, prostate, melanoma, bladder/ureteral, esophageal, gastric, pancreatic, kidney, liver/biliary, uterine, cervical, ovarian, sarcoma. (superficial disease and in situ disease only is excluded)
* Eligible hematologic malignancies include lymphoma any subtype any stage in remission, multiple myeloma in remission, leukemia any subtype in remission.
* Eligible prior cancer treatment modalities include surgery, radiation, chemotherapy, hormonal therapies, immunotherapy, biologic therapies.
* All anti-cancer therapy completed > 6 months prior to enrollment with < 5 years from treatment
* Presence of self-reported fatigue defined by a response of "somewhat, quite a bit, or very much" to the screening question "During the past seven days, did you feel fatigued: Not at all, a little bit, somewhat, quite a bit, very much?"
* Ability to walk without requiring assistance from another individual (use of cane or walker acceptable)
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Unable or unwilling to give informed consent
* Female patients are of childbearing potential, defined as postmenopausal for at least 1 year.
* Prisoners, institutionalized individuals, or others who may be considered vulnerable populations, such as individuals with dementia
* Currently taking warfarin or Coumadin
* Currently taking a steroid medication either regularly or within the last two weeks.
* Patients currently taking medications that are sensitive to substrates or substrates with a narrow therapeutic range for CYP1A2, CYP2C8, CYP2C9, CYP2C19, CYP2D6, CYP3A4, OATP1B1 (Unless willing and able to stop or modify the dosing of the drug) or strong inhibitors or inducers of CYP3A4 (e.g., cyclosporine, tacrolimus, or sirolimus) are excluded, unless medication can be safely held during the following times:
* Immediately before the 1st IP administration (Day 0 or Day 30) until at least 10 hours after the 2nd IP administration (Day 1 or Day 31)
* Immediately before the 3rd IP administration (Day 7 or Day 37) until at least 10 hours after the 4th IP administration (Day 8 or Day 38)
* Subjects taking any of the medications listed in Appendix I may participate if they are otherwise eligible AND the medication can be safely held during the following times: Immediately before the 1st IP administration (Day 0 or Day 30) until at least 10 hours after the 2nd IP administration (Day 1 or Day 31); Immediately before the 3rd IP administration (Day 7 or Day 37) until at least 10 hours after the 4th IP administration (Day 8 or Day 38)
* Drugs listed as part of the exclusion criteria are not permitted during each of the two 2-day courses of treatment with Fisetin. If patients are required to initiate these medications within the 2-day period, they will be removed from the study primarily due to risk of drug-drug interaction.
* Uncontrolled hypertension (systolic >170 OR diastolic >100 mmHg) upon repeated assessments
* Uncontrolled (as per clinical judgement) pleural/pericardial effusions or ascites
* Active malignancy or on-going cancer treatment including oral anti-estrogen therapy, immunotherapy, biologic therapy.
* Men receiving androgen deprivation therapy
* Symptomatic congestive heart failure
* Lung disease requiring oxygen
* End stage renal disease requiring dialysis
* Inability to swallow capsules
* Chronic nausea or diarrhea defined by a frequency of ≥ once per week
* Diagnosis of dementia
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known untreated hypothyroidism
* Allergy to fisetin
* Human immunodeficiency virus infection
* Known active untreated hepatitis B or C infection
* Active invasive fungal infection
* Unwilling to provide informed consent, including consent to access electronic health records
* Judged unsuitable for the trial for any reason by research team
* The following laboratory tests as indicated or as per clinical judgement: Normal organ and marrow function as defined: Hemoglobin <10g/dL, leukocytes <3,000/mcL, absolute neutrophil count <1,500/mcL, platelets <100,000/mcL, total bilirubin above normal institutional limits, AST(SGOT)/ALT(SGPT) >2.5 X institutional upper limit of normal, creatinine clearance <30 mL/min, fasting glucose >300 on day of screening (from plasma or serum)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pittsburgh Fatigability Scale (PFS) | Baseline to Week 2
  10-item PFS score is a measure of perceived fatigability in older adults and can serve as an adjunct to performance-based fatigability measures for identifying older adults at risk of mobility limitation in clinical and research settings. Total score range is 0-50 with higher score indicating greater fatigue.
Change in Pittsburgh Fatigability Scale (PFS) | Baseline to Week 4
  10-item PFS score is a measure of perceived fatigability in older adults and can serve as an adjunct to performance-based fatigability measures for identifying older adults at risk of mobility limitation in clinical and research settings. Total score range is 0-50 with higher score indicating greater fatigue.
Change in Pittsburgh Fatigability Scale (PFS) | Baseline to Week 6
  10-item PFS score is a measure of perceived fatigability in older adults and can serve as an adjunct to performance-based fatigability measures for identifying older adults at risk of mobility limitation in clinical and research settings. Total score range is 0-50 with higher score indicating greater fatigue.
Change in Pittsburgh Fatigability Scale (PFS) | Baseline to Week 12
  10-item PFS score is a measure of perceived fatigability in older adults and can serve as an adjunct to performance-based fatigability measures for identifying older adults at risk of mobility limitation in clinical and research settings. Total score range is 0-50 with higher score indicating greater fatigue.

SECONDARY OUTCOMES:
Change in Patient Reported Outcomes Measurement System (PROMIS) | Baseline to Week 2, Baseline to Week 4, Baseline to Week 6, Baseline to Week 12
  PROMIS Fatigue Short-Form 7a - Item responses are rated on a five-point scale ranging from "never" to "always." Total score range is 5-35 with a higher scores indicating more fatigue.
Change in Pepper Assessment Tool for Disability (PAT-D) | Baseline to Week 2, Baseline to Week 4, Baseline to Week 6
  The (PAT-D) is a 19-item survey to assess domains of physical function in older adults. Responses are made on a five-point Likert scale ranging from "usually did with no difficulty" to "unable to do." Total score range is 19-95 with lower scores indicating better mobility and ability to perform activities of daily and instrumental activities of daily living.
Change in Expanded Short Physical Performance Battery (eSPPB) | Baseline to Week 2, Baseline to Week 4, Baseline to Week 6
  eSPPB is used to objectively assess lower extremity physical function. This validated measure comprises a short walk, narrow walk, repeated chair stands, and balance tests. Total score range is 0-12 with higher scores indicating better physical performance. Lower scores on the eSPPB have been associated with increased risk of disability, hospitalization and worse survival among older adults with and without cancer.
Change in 6-minute Walk Distance | Baseline to Week 2, Baseline to Week 4, Baseline to Week 6
  Distance participant is able to walk in 6-minute will be measured. The 6-minute walk accurately assesses submaximal exercise capacity and is an independent predictor of mortality and is correlated with peak V02 testing.
Change in Fried Frailty Phenotype Score | Baseline to Week 2, Baseline to Week 4, Baseline to Week 6
  Frailty score is calculated using the Frailty Index Calculation form. Score range is 0-5 with a higher score indicating frailty.
Change in Longitudinal Aging Study Amsterdam (LASA) Sedentary Behavior Questionnaire | Baseline to Week 2, Baseline to Week 4, Baseline to Week 6
  10-item questionnaire used to measure sedentary behavior. The average time per 24 hours spent on each individual sedentary activity will be recorded in hours and/or minutes. This will be done for an average weekday as well as for an average weekend day. Ranges from 0-24 hours with a higher score indicating more sedentary behavior.
Change in PROMIS Global Health Short Form | Baseline to Week 2, Baseline to Week 4, Baseline to Week 6
  PROMIS Global Health Short Form is a 10-item instrument assesses the extent to which patients experience problems with fatigue over the past 7 days using a 5-point Likert scale. The fatigue subscale provides a raw score, ranging from 4 to 20. Raw scores are converted to T-scores using the PROMIS conversion tables. Higher scores reflect greater fatigue.
Medication Adherence Rate | Week 2, Week 5
  Empty bottles from home will be returned. The number of pills taken is calculated by subtracting the count of the number of pills remaining from the total number of pills dispensed. The drug adherence rate is then calculated by dividing the number of pills taken by the number of pills they were supposed to take.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kritchevsky, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist Hospital, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No